CLINICAL TRIAL: NCT05776121
Title: A Multiple Ascending Doses Study of ZB001 in Chinese Patients With Thyroid-Associated Ophthalmopathy
Brief Title: Study of ZB001 in Chinese Patients With Thyroid Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZB001-01-002
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZB001 for injection (Experimental): Treat different dose cohorts with four intravenous injections of ZB001
  Interventions: Drug: ZB001 for injection

INTERVENTIONS:
Drug: ZB001 for injection — Dose Cohort1 (3 mg/kg) ZB001 four IV injections
Drug: ZB001 for injection — Dose Cohort2 (10 mg/kg) ZB001 four IV injections

SUMMARY:
The investigational drug, ZB001 is a humanized IgG1κ monoclonal antibody targeting human IGF-1R. The study is designed to evaluate the efficacy, safety, tolerability, and pharmacokinetics（PK）/pharmacodynamics (PD) profile of ZB001 in Chinese patients with Thyroid Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, 18 years of age or older
2. Clinical diagnosis of Graves' ophthalmopathy and CAS evaluation of eyes under study ≥ 4 points (7 points in total)
3. Moderate-to-severe active thyroid-associated ophthalmopathy (i.e., severely affects daily life): exophthalmos extent is ≥18.6 mm, or progressive exophthalmos (≥3 mm greater than the previous exophthalmos record per the investigator); accompanied by at least one of the following symptoms: eyelid retraction ≥ 2 mm; moderate or severe soft tissue involvement (conjunctival congestion, edema, periorbital congestion or edema); non-persistent or persistent diplopia
4. Before Screening, evidence of eye symptoms or signs related to thyroid-associated ophthalmopathy in medical records for ≤1 year
5. Thyroid function normal, or only mild hyperthyroidism or hypothyroidism, defined as free thyroxine (FT4) ）and free triiodothyronine (FT3) levels within 0.5-1.5 times the normal range at Screening. Efforts have been made to correct any mild hypothyroidism or hyperthyroidism in a timely manner and try to maintain normal thyroid function throughout the study. Thyroidectomy is not an exclusion.
6. If the patient is a female of childbearing potential (including a female with menopause < 1 year, amenorrhea < 1 year, or without surgical sterilization), the pregnancy test result will be negative at Screening. Such patients must agree to use the effective birth control methods described in the relevant protocol section (Section 9.2 Contraception and Pregnancy) at least one complete menstrual cycle before the first dose of the study drug, and continue to use contraception methods for 100 days after the last dose
7. Male patients must be surgically sterilized for at least 6 weeks or agree to use the effective birth control methods described in the relevant protocol section (Section 9.2 Contraception and Pregnancy) before the first dose of the study drug and within 100 days after the last dose

Exclusion Criteria:

1. In the past 6 months, due to optic neuropathy, new visual field defect or color defect secondary to optic nerve involvement, the best corrected visual acuity of the study eye decreased, defined as the result of standardized visual acuity chart decreased ≥ 0.2
2. Corneal involvement of the study eye, and no improvement after medical interventions
3. CAS decreased ≥ 2 points from Screening Assessment to Day -1
4. The exophthalmos extent of the study eye ≥ 2 mm from Screening Assessment to Day -1
5. The study eye previously received orbital radiotherapy or surgery due to thyroid-associated ophthalmopathy
6. Known history of clinically significant ear disease, ear surgery or hearing loss
7. Inflammatory bowel disease (e.g., biopsy-proven or clinical evidence of inflammatory bowel disease)
8. Cumulative use of glucocorticoid equivalent to ≥ 1g methylprednisolone as thyroid-associated ophthalmopathy treatment (A lower cumulative dose [<1g] of glucocorticoid used before Screening, or hormone eye drops withdrawn for ≥ 6 weeks before Screening, is allowed for inclusion)
9. Received any doses of oral corticosteroids to treat diseases other than thyroid-associated ophthalmopathy within 4 weeks before Screening (local application is allowed for inclusion)
10. Pregnant or lactating females
11. Smokers (≥ 5 cigarettes/day) or former smokers (≥ 5 cigarettes/day) quit within 6 months before enrollment in the study
12. Any vaccination planned during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events, Serious Adverse Events, and Laboratory Evaluations as assessed by CTCAE v5.0 | through study completion, up to 169 days
The exophthalmos response rates of study eye at Week 6 and Week 12 (defined as the proportion of patients whose exophthalmos measured by Hertel exophthalmos meter decreased ≥ 2mm from baseline) | At week6 and week 12

SECONDARY OUTCOMES:
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Exophthalmos measured by MRI/CT scan | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Orbital fat volume measured by MRI/CT scan | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Extraocular eye muscle volume measured by MRI/CT scan | At week6, week 12 and week24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Facial fat volume measured by MRI/CT scan | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Digital and manual measurement of palpebral fissure height | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Exotropia deviation measurement | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Subjective diplopia score. The range of score is from 0-3. The lower score means the better outcome. | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Best corrected visual acuity | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Intraocular pressure | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Clinical Activity Score (CAS) . The range of score is from 0-7. The lower score means the better outcome | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Graves ophthalmopathy - Quality of Life (QoL). The range of score is from 0-100. The higher change of quality of life means the better outcome. | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Graves ophthalmopathy - Visual function QOL. The range of score is from 0-100. The higher change of quality of life means the better outcome. | At week6, week 12 and week 24
Change from baseline in the study eye at Week 6, Week 12 and Week 24 of Graves ophthalmopathy - Social Function QoL. The range of score is from 0-100.The higher change of quality of life means the better outcome. | At week6, week 12 and week 24
Serum ZB001 antidrug antibody (ADA) titers | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  antidrug antibody (ADA) titers of ZB001
Serum IGF-1 concentrations in the blood over time | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
Maximum observed concentration (Cmax) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Time to measured peak concentration (Tmax) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Area under the concentration-time curve from time 0 to the last timepoint with measurable concentration (AUClast) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Area under the concentration-time curve extrapolated to infinity (AUCinf) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Area under the concentration-time curve over a dosing interval (AUCtau) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
half life (t1/2) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Systemic clearance (CL) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
Steady State Volume of Distribution (Vss) | Before and after drug administration, performed according to the protocol visit time specified in the plan, up to 169 days
  Pharmacokinetics
The exophthalmos response rates of study eye at Week 24 (defined as the proportion of patients whose exophthalmos measured by Hertel exophthalmos meter decreased ≥ 2mm from baseline) | At week6 and week 12

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing
  - Peking University Third Hospital, Beijing
  - Third Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Chongqing Aier General Hospital, Chongqing
  - The Second Hosptial of Dalian Medical University, Dalian
  - The Second Hosptial of Anhui Medical University, Hefei
  - Affiliated Eye Hospital of Nanchang University, Nanchang